CLINICAL TRIAL: NCT05849935
Title: A Study to Establish a Reference Range for abioSCOPE® Device With the PSP Assay in a Generally Healthy Adult Population
Brief Title: abioSCOPE PSP Reference Range Study; Extension of AB-PSP-003
Acronym: AB-PSP-007
Status: Completed | Type: Observational
Sponsor: Abionic SA (Industry)
Collaborators: Avania (Industry)
Responsible Party: Sponsor
Other Study IDs: AB-PSP-007
Record Dates: First submitted 2023-04-28; First posted 2023-05-09 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-07

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: abioSCOPE — The abioSCOPE device with the PSP assay is intended to be indicated for ICU admitted patients at risk of developing sepsis. Results of abioSCOPE PSP assay may aid to identify sepsis in critically ill patients, together with all other clinical assessment and laboratory findings.

SUMMARY:
This is a monocentric, prospective, biomarker-result-blinded observational study evaluating immunoassay measurements of pancreatic stone protein (PSP) performed on Abionic's abioSCOPE device with the PSP assay on generally healthy adults representative of the US population.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged ≥ 18 years.
2. Apparently healthy as determined by a subject questionnaire.

Exclusion Criteria:

1. Current diagnosis, or history, of any underlying major medical condition determined by the investigator, including but not limited to

   1. Renal disease
   2. Stoke
   3. Liver disease
   4. Pancreatic disease (including diabetes)
   5. HIV AIDS
   6. Receiving antibiotic therapy
   7. Suspected infection
   8. Immunosuppression
2. Underwent procedures related to sepsis, or diagnosed with sepsis, within the last 12 months.
3. Current diagnosis of uncontrolled diabetes.
4. Diagnosis of bacterial, fungal, or malaria infection within the last 3 months that required antimicrobial treatment.
5. Experienced severe trauma, surgery, cardiac arrest, or severe burn within the previous 3 months requiring medical care.
6. Diagnosis and/or treatment of cancer within the last 12 months.
7. Received immunosuppressive therapy.
8. Hospitalization for more than 24 hours within the last month.
9. Reported as currently pregnant or nursing a child
10. Unable or unwilling to provide the required blood sample for testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult healthy population
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2023-07-17 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
To determine the reference range intervals of PSP values measured using abioSCOPE device with the PSP assay in a generally healthy population representative of the US population. | through study completion, an average of 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sundance Clinical, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No